CLINICAL TRIAL: NCT05885789
Title: Improvement of Laryngoscopic View by Bed-up-head-elevated Position During Tracheal Intubation in Paediatric Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Malaya (Other)
Responsible Party: Principal Investigator, Kim Bao Zhen, Principal investigator, University of Malaya
Other Study IDs: BUHE in paediatric
Record Dates: First submitted 2023-05-22; First posted 2023-06-02 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-06

CONDITIONS: Paediatric Airway Management
Keywords: Paediatric; Intubation; Laryngoscopy; Head position; BUHE
MeSH Terms: interventions — Intubation; Patient Positioning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Paediatric patients
  Interventions: Procedure: Intubation in Bed-Up-Head-Elevated (BUHE) position

INTERVENTIONS:
Procedure: Intubation in Bed-Up-Head-Elevated (BUHE) position — Comparing laryngoscopic view in paediatric patients during sniffing position and BUHE position

SUMMARY:
The goal of this prospective observational study is to learn about improvement of laryngoscopic view by Bed-Up-Head-Elevated (BUHE) during tracheal intubation in paediatric patients. The main question it aims to answer is:

1. Does BUHE position improve laryngoscopic view during paediatric intubation?

Participants age 3-12 year-old going for elective surgery under general anaesthesia requiring tracheal intubation will undergo laryngoscopic twice, first in sniffing position (SP) and second during BUHE position.

POGO score during each laryngoscope will be compared. Additionally, ease of handling of laryngoscope during each position will be assessed.

DETAILED DESCRIPTION:
This is a prospective observational study comparing POGO score during tracheal intubation in SP and BUHE position in paediatric patients aged 3 to 12 years who will undergo elective surgery under general anaesthesia requiring tracheal intubation. The first POGO score will be obtained during SP followed by second POGO score during BUHE position and the difference in POGO score before and after BUHE position will be recorded to learn the improvement in POGO score during BUHE position.

The objective of this study is to learn the improvement of laryngeal view in tracheal intubation after BUHE position in paediatric patients of age 3 to 12 years. Investigators hypothesised that laryngeal view in tracheal intubation improves after BUHE position compared to sniffing position.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to 12 years
* Elective surgery under general anaesthesia requiring tracheal intubation

Exclusion Criteria:

* Parents' / Guardian's refusal
* Known case of difficult airway or airway malformation or airway obstruction
* Patients with respiratory or cardiovascular disease
* Patients requiring rapid sequence induction
* Recent Upper Respiratory Tract Infection (URTI) of 2 weeks

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Paediatric patients age 3-12 year-old undergoing elective surgery under general anaesthesia requiring tracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Percentage of Glottic Opening (POGO) score after BUHE position | Immediate during procedure
  Compare change in Percentage of Glottic Opening (POGO) score in sniffing position (SP) and after BUHE position. The POGO score is expressed as a percentage of glottis exposure in the laryngoscopy view, which is expressed as 100% for a fully exposed glottis, from the anterior commissure of the vocal cords to the inter-arytenoid notch. POGO score of 0% corresponds to no visualisation of laryngeal structure.

SECONDARY OUTCOMES:
Ease of handling of laryngoscope | Immediate during procedure
  assessed based on a scale of 0 to 10, 0 being the most difficult and uncomfortable handling and 10 being the easiest and most comfortable handling

CONTACTS AND LOCATIONS:
Overall Officials: Bao Zhen Dr. Kim, MD, Principal Investigator — University of Malaya Medical Center
Locations (1):
- University of Malaya Medical Center, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Study Protocol Statistical Analysis Plan (SAP) Clinical Study Report (CSR)

REFERENCES:
- [Background] Karsli C. Managing the challenging pediatric airway: Continuing Professional Development. Can J Anaesth. 2015 Sep;62(9):1000-16. doi: 10.1007/s12630-015-0423-y. Epub 2015 Aug 5. PMID 26243378
- [Background] Schmidt AR, Weiss M, Engelhardt T. The paediatric airway: basic principles and current developments. Eur J Anaesthesiol. 2014 Jun;31(6):293-9. doi: 10.1097/EJA.0000000000000023. PMID 24247412
- [Background] Holm-Knudsen RJ, Rasmussen LS. Paediatric airway management: basic aspects. Acta Anaesthesiol Scand. 2009 Jan;53(1):1-9. doi: 10.1111/j.1399-6576.2008.01794.x. PMID 19128325
- [Background] Vialet R, Nau A. Effect of head posture on pediatric oropharyngeal structures: implications for airway management in infants and children. Curr Opin Anaesthesiol. 2009 Jun;22(3):396-9. doi: 10.1097/aco.0b013e3283294cc7. PMID 19434789
- [Background] Kim EH, Ji SH, Song IK, Lee JH, Kim JT, Kim HS. Simple method for obtaining the optimal laryngoscopic view in children: A prospective observational study. Am J Emerg Med. 2017 Jun;35(6):867-870. doi: 10.1016/j.ajem.2017.01.048. Epub 2017 Jan 24. PMID 28139308
- [Background] Ahn JH, Kim D, Gil NS, Son YH, Seong BG, Jeong JS. Improvement of laryngoscopic view by hand-assisted elevation and caudad traction of the shoulder during tracheal intubation in pediatric patients. Sci Rep. 2019 Feb 4;9(1):1174. doi: 10.1038/s41598-018-37770-6. PMID 30718623
- [Background] Lee BJ, Kang JM, Kim DO. Laryngeal exposure during laryngoscopy is better in the 25 degrees back-up position than in the supine position. Br J Anaesth. 2007 Oct;99(4):581-6. doi: 10.1093/bja/aem095. Epub 2007 Jul 4. PMID 17611252
- [Background] Black AE, Flynn PE, Smith HL, Thomas ML, Wilkinson KA; Association of Pediatric Anaesthetists of Great Britain and Ireland. Development of a guideline for the management of the unanticipated difficult airway in pediatric practice. Paediatr Anaesth. 2015 Apr;25(4):346-62. doi: 10.1111/pan.12615. Epub 2015 Feb 16. PMID 25684039
- [Result] Tsan SEH, Lim SM, Abidin MFZ, Ganesh S, Wang CY. Comparison of Macintosh Laryngoscopy in Bed-up-Head-Elevated Position With GlideScope Laryngoscopy: A Randomized, Controlled, Noninferiority Trial. Anesth Analg. 2020 Jul;131(1):210-219. doi: 10.1213/ANE.0000000000004349. PMID 31348051